CLINICAL TRIAL: NCT00272909
Title: A Phase IIb Randomized, Double-blind, Placebo-Controlled, Group-Sequential, Multicenter, Dose Finding Study of the Safety and Efficacy of SUN N4057 (Piclozotan) Administered for 72 Hours by Continuous Intravenous Infusion in Subjects With Acute Ischemic Stroke and Measurable Penumbra on MRI
Brief Title: Efficacy of SUN N4057 in Subjects With Acute Ischemic Stroke and Measurable Penumbra on Magnetic Resonance Imaging (MRI)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Ron Corey, PhD, MBA Executive Director, Clinical and Project Management, Asubio Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-103
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Stroke
Keywords: Acute Ischemic Stroke; 9-Hour window MRI; Serotonin receptor agonist
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Piclozotan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): piclozotan IV infusion, low dose, for 72 hours.
  Interventions: Drug: piclozotan low dose
- 2 (Experimental): piclozotan IV infusion, high dose, for 72 hours.
  Interventions: Drug: piclozotan high dose
- 3 (Placebo Comparator): placebo (normal saline) IV infusion, for 72 hours.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: piclozotan low dose — Continuous IV infusion over a period of up to 72 hours of piclozotan
  Arms: 1
Drug: placebo — Continuous IV infusion over a period of up to 72 hours of placebo.
  Arms: 3
Drug: piclozotan high dose — Continuous IV infusion over a period of up to 72 hours of piclozotan
  Arms: 2

SUMMARY:
This research study is designed to evaluate the safety, tolerability, and efficacy of SUN N4057 (piclozotan) in subjects with acute ischemic stroke within 9 hours of the onset of symptoms.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the efficacy of a 72 hour infusion of SUN N4057 (piclozotan) in subjects with clinical findings of an acute ischemic stroke and a magnetic resonance imaging (MRI) demonstrating a measurable penumbra (perfusion-weighted imaging [PWI] minus diffusion-weighted imaging [DWI] volume). Efficacy will be determined by comparing the proportion of subjects with no growth in stroke lesion volume as assessed by DWI at Screening to stroke lesion volume assessed by FLAIR (fluid-attenuated inversion recovery) on Day 28 in the piclozotan group versus the placebo group.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

* Males or females >= 18 and <= 85 years of age at randomization. Female subjects must be either:

  * Surgically sterile;
  * Postmenopausal for at least 1 year; or
  * Non-pregnant, confirmed by a serum pregnancy test, and using a method of birth control that is acceptable to the investigator.
* Neurological examination demonstrating localizing cortical signs
* Receipt of study drug less than 6 hours (50% of subjects) or between 6 and 9 hours, inclusive, (50% of subjects) after the onset of symptoms (for un-witnessed stroke, last time seen in normal state or at bedtime for un-witnessed stroke during sleep)
* Signed informed consent from subject or legally acceptable representative
* NIHSS score of 6 - 22, inclusive, or at least 2 on the aphasia item of the NIHSS with a location of MRI findings consistent with aphasia

MRI-determined inclusion criteria:

* Acute ischemic stroke with substantial cortical involvement in the middle cerebral artery (MCA) distribution, as verified by the Screening DWI abnormality and/or Screening PWI abnormality. (Note: white matter involvement, in addition to cortex, is not an exclusion.)

Exclusion Criteria:

General exclusion criteria:

* Two or more of the following:

  * Reduced level of consciousness (score >= 2 on NIHSS Q1a)
  * Forced eye deviation or total gaze paresis (score of 2 on NIHSS Q2)
  * Dense hemiplegia (no movement) of upper and lower extremities (score of 4 on NIHSS Q5 regarding motor arm and a score of 4 on NIHSS Q6 regarding motor leg)
* Pre-stroke modified Rankin score >= 2 at Screening
* Rapid neurological improvement from Screening up to the start of drug infusion
* Persistent systolic blood pressure (SBP) > 220 mmHg and/or diastolic blood pressure (DBP) > 120 mmHg (confirmed by at least three readings taken at least 3 minutes apart) prior to randomization. If subsequent readings are consistently below these levels, either spontaneously or following mild antihypertensive therapy, subject may be enrolled.

MRI-determined exclusion criteria:

* Intracranial hemorrhage as verified by Screening MRI. (Note: intracranial hemorrhage on pre-screen computerized tomography [CT] scan also excludes subject.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-09; Primary Completion 2006-10 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Improvement in MRI | 28 days

SECONDARY OUTCOMES:
The change in stroke lesion volume from Screening to day 28 | 28 days
Clinical outcomes at Days 28 and 90 using the individual clinical scales (Modified Rankin Scale, Barthel Index, and National Institutes of Health Stroke Scale [NIHSS]). | Days 28 and 90
To assess the safety and tolerability of SUN N4057 (piclozotan) in subjects with acute stroke. | Days 28, 60 and 90

CONTACTS AND LOCATIONS:
Locations (47):
- United States (25):
  - UCLA Stroke Network, Los Angeles, California
  - San Francisco Clinical Research Center, San Francisco, California
  - The Stroke Center at Hartford Hospital, Hartford, Connecticut
  - Lakeland Regional Medical Center, Lakeland, Florida
  - OCALA Neurodiagnostic Center, Ocala, Florida
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Ruan Neurology Clinic and Clinical Research Center, Des Moines, Iowa
  - Via Christi Regional Medical Center, Wichita, Kansas
  - University of Kentucky, Sanders Brown Center on Aging/Stroke Program, Lexington, Kentucky
  - University of Massachusetts, Memorial Health Center, Department of Neurology, Worcester, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Michigan State University, Sparrow Health System, East Lansing, Michigan
  - St. Luke's Hospital, Kansas City, Missouri
  - Advance Neurology Specialists, Great Falls, Montana
  - St. Francis Medical Center, Trenton, New Jersey
  - SUNY at Stony Brook, University Hospital at Stony Brook, Stony Brook, New York
  - Moses Cone Hospital, Greensboro, North Carolina
  - Clinical Research Center of Winston-Salem, Winston-Salem, North Carolina
  - Summa Health System Neurology and Neuroscience Associates, Akron, Ohio
  - Chattanooga Neurology Associates, Chattanooga, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - The Methodist Hospital Neurological Institute, Houston, Texas
  - INOVA Research Center, Falls Church, Virginia
  - Charleston Area Medical Center Health Education and Research Institute, Charleston, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (3):
  - General Hospital Middelheim, Dept. of Neurology, Antwerp
  - Hopital Erasme - Dept. of Neurology, Universite Libre de Bruxelles, Brussels
  - Uz Gasthuisberg, Neurology, Leuven
- Germany (4):
  - Universitatsklinikum Essen, Department of Neurology, Essen
  - Neurologische Universitatsklinik und Poliklinik - Neurzentrum, Freiburg im Breisgau
  - Universitatsklinikum Leipzig Aor, Klinik And Poliklinok Fur Neurologie, Leipzig
  - Neurologische Klinik, Klinikum Rechts Der Isar Der Tu Munchen, München
- Israel (6):
  - Soroka University Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah University Hospital, Jerusalem
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Center, Zrifin
- Poland (3):
  - Centralny Szpital Kliniczny, Katowice
  - Collegium Medicum Jegiellonian University, Krakow
  - Military Institute of Medicine, Warsaw
- South Africa (3):
  - St Augustines Hospital, Durban
  - Vergelegen Medi-Clinic, Somerset West
  - Sunninghill Hospital Cnr., Sunninghill
- Spain (3):
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - University Hospital of Girona Dr. Josep Trueta, Neurology Department, Girona
  - Hospitales Universitarios Virgen Del Rocio, Seville